CLINICAL TRIAL: NCT03964337
Title: A Phase II, Open-Label Randomized Study of Immediate Prostatectomy vs. Cabozantinib Followed by Prostatectomy in Men With High-Risk Prostate Cancer (SPARC)
Brief Title: Immediate Prostatectomy vs. Cabozantinib Followed by Prostatectomy in Men With High-Risk Prostate Cancer
Acronym: SPARC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual.
Sponsor: Duke University (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00101042
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer; Prostate Cancer Adenocarcinoma; Non-Metastatic
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cabozantinib Followed by Prostatectomy (Arm A) (Experimental): Experimental group will received cabozantinib for 4 weeks, followed by a 2 week drug washout before a prostatectomy.
  Interventions: Drug: Cabozantinib; Procedure: Radical Prostatectomy
- Immediate Prostatectomy (Arm B) (Active Comparator): Control group will receive an immediate prostatectomy.
  Interventions: Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib 40 mg by mouth daily for 4 weeks.
  Other Names: Cabometyx
  Arms: Cabozantinib Followed by Prostatectomy (Arm A)
Procedure: Radical Prostatectomy — Radical prostatectomy as part of routine medical care.

SUMMARY:
This is a prospective, randomized, open-label, phase II trial of cabozantinib in subjects with untreated, high risk prostate cancer undergoing radical prostatectomy. This multicenter study will enroll 30 subjects. Duke is the lead site for this trial. There will be a second site selected TBD.

Patients will be assigned (first 9 subjects only) or randomized 2:1 to either: (1) cabozantinib 40 mg by mouth daily for 4 weeks, followed by a 2 week drug washout period before prostatectomy (n = 20), or (2) immediate prostatectomy within 12 weeks of registration (n = 10). The first 9 subjects (6 subjects assigned to cabozantinib treatment, 3 subjects assigned to immediate prostatectomy) will constitute the Safety Lead-In Cohort, which will be only accrued at Duke. After six subjects have received cabozantinib and completed the 57-85 day safety visit without triggering a stopping rule, subjects may be accrued at the ex-Duke site.

The primary goal is to compare pathologic apoptotic indices (cleaved caspase-3) in prostatectomy specimens from patients who undergo immediate prostatectomy (controls) versus those who receive with cabozantinib followed by prostatectomy. The secondary objective is to conduct immune phenotypic profiling on the peripheral blood and tumor microenvironment in prostatectomy specimens from both groups. A statistical analysis will be used to compare the apoptotic indices between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age ≥ 18 years old.
2. ECOG performance status of 0 or 1
3. Histologic evidence of adenocarcinoma of the prostate who are deemed candidates for curative radical prostatectomy.
4. Planned robotic or laparoscopic prostatectomy technique.
5. Low risk for conversion to open prostatectomy, in the opinion of the treating surgeon.
6. Intermediate-high or high risk, clinically localized disease by the following criteria:

   * Prostate cancer in at least 2 cores with a Gleason score ≥ 7 (4+3 or 3+4) in at least 1 of those cores.
   * No definite evidence of metastasis, in the opinion of the investigator.
7. Adequate organ function as defined by the following criteria within 14 days prior to first dose of study treatment:

   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3 x local laboratory upper limit of normal (ULN)
   * Total serum bilirubin ≤1.5 x ULN, (for subjects with Gilbert's disease ≤ 3 x ULN)
   * Absolute neutrophil count (ANC) ≥1500/L without granulocyte colony-stimulating factor support.
   * White blood cell count ≥ 2500/mm3
   * Serum albumin ≥ 2.8 g/dl
   * Platelets ≥100,000/mm3
   * Hemoglobin ≥9.0 g/dL
   * Serum calcium ≤12.0 mg/dL
   * Serum creatinine ≤ 2.0 x ULN or calculated creatinine clearance ≥ 30mL/min.
   * Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol).
8. Written Authorization for Use and Release of Health and Research Study Information (HIPAA authorization per institutional requirements)
9. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
10. Willing/able to adhere to the prohibitions and restrictions specified in this protocol.
11. Agrees to use a condom (even men with vasectomies) and another effective method of birth control if subject is having sex with a woman who is pregnant or a woman of childbearing potential while on study drug and for 4 months following the last dose of study drug.

Exclusion Criteria:

1. Prior treatment for prostate cancer.
2. Major surgery or radiation therapy within 4 weeks of Day 1 on study.
3. Planned radiation therapy until at least 4 weeks after prostatectomy.
4. NCI CTCAE v4.0 grade 3 hemorrhage within 4 weeks of Day 1 on study.
5. Prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥ 1.3 x the laboratory ULN within 14 days before Day 1 on study (Arm A subjects only) or within 14 days of the completion of screening (Arm B subjects only).
6. Concomitant anticoagulation with oral anticoagulants (e.g., warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel). However, low-dose aspirin for cardio protection is allowed (per local applicable guidelines).
7. History of or known metastatic prostate cancer.
8. QTcf interval > 500 msec on baseline EKG.
9. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   a. Cardiovascular disorders:

   i. Symptomatic congestive heart failure (CHF) New York Heart Association Class 3 or 4, unstable angina pectoris, ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2. coronary/peripheral artery bypass graft (CABG), within 6 months prior to screening.

   ii. Stroke (including transient ischemic attack [TIA]), cerebrovascular accident (CVA), myocardial infarction (MI), or other ischemic event, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism (PE)) within 6 months prior to screening.

   b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

   i. Evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.

   ii. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose.

   Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose.

   c. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose.

   d. Serious non-healing wound/ulcer/bone fracture. e. Other clinically significant disorders that would preclude safe study participation.
10. Hypertension that cannot be controlled by medications (>140/90 mm Hg despite optimal medical therapy).
11. Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
12. Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
13. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
14. Inability to swallow tablets.
15. Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harrison, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study accrual was discontinued prior to enrolling any participants in the control arm (Immediate Prostatectomy, Arm B).
Period: Overall Study
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study accrual was discontinued prior to enrolling any participants in the control arm (Immediate Prostatectomy, Arm B).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B) | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.47 (8.40) |  | 62.47 (8.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 3 |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Apoptotic Index in Prostatectomy Specimens From Patients Who Undergo Immediate Prostatectomy (Arm B) Versus Those Treated With Cabozantinib Followed by Prostatectomy (Arm A)
Description: Apoptotic index as measured by cleaved caspase-3 levels in tumor tissue
Time Frame: At prostatectomy (Arm A: Day 43, Arm B: Day 1)
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Immune Phenotyping of Myeloid-derived Suppressor Cells (MDSCs)
Description: Percentage of MDSCs in peripheral blood and tumor tissue
Time Frame: Arm A: Screening, Day 29, Day 43, Day 57-85; Arm B: Screening, Day 1
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Immune Phenotyping of Neutrophils
Description: Percentage of neutrophils in peripheral blood and tumor tissue
Time Frame: Arm A: Screening, Day 29, Day 43, Day 57-85; Arm B: Screening, Day 1
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Immune Phenotyping of M1 Macrophages
Description: Percentage of M1 macrophages in peripheral blood and tumor tissue
Time Frame: Arm A: Screening, Day 29, Day 43, Day 57-85; Arm B: Screening, Day 1
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Immune Phenotyping of M2 Macrophages
Description: Percentage of M2 macrophages in peripheral blood and tumor tissue
Time Frame: Arm A: Screening, Day 29, Day 43, Day 57-85; Arm B: Screening, Day 1
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Immunohistochemical (IHC) Analysis of CD8+
Description: Percentage of CD8+ positive cells in tumor tissue
Time Frame: At prostatectomy (Arm A: Day 43, Arm B: Day 1)
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Immunohistochemical (IHC) Analysis of Programmed Death Ligand-1 (PD-L1)
Description: Percentage of PD-L1 positive cells in tumor tissue
Time Frame: At prostatectomy (Arm A: Day 43, Arm B: Day 1)
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Immunohistochemical (IHC) Analysis of Cytotoxic T-lymphocyte-associated Protein 4 (CTLA-4)
Description: Percentage of CTLA-4 positive cells in tumor tissue
Time Frame: At prostatectomy (Arm A: Day 43, Arm B: Day 1)
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Immunohistochemical (IHC) Analysis of Interleukin-1 Receptor Antagonist (IL-1RA)
Description: Percentage of IL-1RA positive cells in tumor tissue
Time Frame: At prostatectomy (Arm A: Day 43, Arm B: Day 1)
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Description of the Neutrophil Chemotactic Factor CXCL12
Description: Percentage of neutrophil chemotactic factor CXCL12 positive cells in tumor tissue
Time Frame: At prostatectomy (Arm A: Day 43, Arm B: Day 1)
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Description of the Neutrophil Chemotactic Factor HMGB1
Description: Percentage of neutrophil chemotactic factor HMGB1 positive cells in tumor tissue
Time Frame: At prostatectomy (Arm A: Day 43, Arm B: Day 1)
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Description of the MDSC-promoting Cytokine CCL5
Description: Percentage of MDSC-promoting cytokine CCL5 positive cells in tumor tissue
Time Frame: At prostatectomy (Arm A: Day 43, Arm B: Day 1)
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Description of the MDSC-promoting Cytokine CCL12
Description: Percentage of MDSC-promoting cytokine CCL12 positive cells in tumor tissue
Time Frame: At prostatectomy (Arm A: Day 43, Arm B: Day 1)
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Description of the MDSC-promoting Cytokine CD40
Description: Percentage of MDSC-promoting cytokine CD40 cells in tumor tissue
Time Frame: At prostatectomy (Arm A: Day 43, Arm B: Day 1)
Population: Data not collected.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Per the protocol, AEs are collected from the first dose of study drug (Day 0) through 30 days after the decision to discontinue study treatment (Day 57).
Description: Study accrual was discontinued prior to enrolling any participants in the control arm (Immediate Prostatectomy, Arm B). AEs were predominantly collected at protocol required study visits. The study coordinator would ask the subject about their health and any side effects they experienced. The investigator would perform a physical exam. Blood was collected for safety labs.
Arm/Group | Cabozantinib Followed by Prostatectomy (Arm A) | Immediate Prostatectomy (Arm B)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib Followed by Prostatectomy (Arm A) (N=3) | Immediate Prostatectomy (Arm B) (N=0)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Investigations - Other (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hair color changes (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study accrual was discontinued prior to enrolling any participants in the control arm (Immediate Prostatectomy, Arm B).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT03964337/Prot_SAP_000.pdf